CLINICAL TRIAL: NCT00001459
Title: Tomographic Myocardial Wall Motion Analysis in Patients With Myocardial Ischemia and in Normal Subjects
Brief Title: Analysis of Heart Muscle Function in Patients With Heart Disease and Normal Volunteers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950048; 95-H-0048
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Cardiomyopathy, Hypertrophic; Coronary Disease; Healthy; Myocardial Ischemia; Syndrome X
Keywords: Gated Blood Pool; SPECT Scan; Coronary Artery Disease; Hypertrophic Cardiomyopathy; Microvascular Angina
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Coronary Disease; Myocardial Ischemia; Microvascular Angina; Coronary Artery Disease

SUMMARY:
Myocardial ischemia is a heart condition in which not enough blood supply and oxygen reaches the heart muscle. Damage to the major blood vessels of the heart (coronary artery disease), minor blood vessels of the heart (microvascular heart disease), or damage to the heart muscle (hypertrophic cardiomyopathy) can cause myocardial ischemia. Any of theses three conditions can cause patients to experience chest pain and other symptoms as well as cause the heart to function improperly.

In order to detect myocardial ischemia researchers can use tests to measure the movement of the walls of the heart. Walls receiving inadequate supplies of blood often move less and occasionally move in the opposite direction. Some of the tests may require patients to receive injections of radioactive tracers. The radioactive material acts to enhance 3 dimensional pictures of the heart and helps to identify areas of ischemia.

The purpose of this study is to determine whether 3-dimensional imaging (tomography) with radioactive tracers can provide more important information about heart wall function than routine diagnostic tests.

DETAILED DESCRIPTION:
We propose to assess regional myocardial function using gated blood pool imaging acquired by a tomographic technique at rest and during stress in patients with myocardial ischemia (coronary artery disease, hypertrophic cardiomyopathy and microvascular angina). Gender differences in response to exercise and pharmacologic stress will also be evaluated. Normal subjects will be studied in order to establish a control database. Current methods of gated blood pool studies use planar imaging, with its attendant limitations; poor resolution and inadequate separation of the myocardial segments, only one view assessed during exercise and superimposition of overlying structures. Tomographic imaging has the advantages of reconstructing 3-dimensional data of the entire heart with the ability to improve segmental resolution and separate overlapping structures, potentially resulting in increased sensitivity and specificity for detection of disease.

The role of pharmacologic stress will be assessed by comparison with exercise stress, in order to validate its use in subjects unable to exercise and identify gender related differences. Quantitative measures of regional wall motion obtained from tomography will be compared to regions of prior myocardial infarction (if present), and with other modalities for evaluating cardiac structure and function. The diagnostic and prognostic value of tomographic wall motion analysis will be studied in patients with myocardial ischemia, with special emphasis on correlation between physiologic variables of coronary blood flow and metabolic function.

ELIGIBILITY:
Patients with known coronary artery disease (obstruction of greater than or equal to 50% in at least one major coronary artery).

Patients with hypertrophic cardiomyopathy.

Patients with microvascular angina.

No unstable angina.

No hepatic or renal failure.

Infective endocarditis

No primary valvular disease.

No congenital heart disease.

No pregnant or breast feeding women.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1995-01; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Faber TL, Stokely EM, Templeton GH, Akers MS, Parkey RW, Corbett JR. Quantification of three-dimensional left ventricular segmental wall motion and volumes from gated tomographic radionuclide ventriculograms. J Nucl Med. 1989 May;30(5):638-49. PMID 2785584
- [Background] Corbett JR, Jansen DE, Lewis SE, Gabliani GI, Nicod P, Filipchuk NG, Redish GA, Akers MS, Wolfe CL, Rellas JS, et al. Tomographic gated blood pool radionuclide ventriculography: analysis of wall motion and left ventricular volumes in patients with coronary artery disease. J Am Coll Cardiol. 1985 Aug;6(2):349-58. doi: 10.1016/s0735-1097(85)80171-6. PMID 2991357
- [Background] Borer JS, Kent KM, Bacharach SL, Green MV, Rosing DR, Seides SF, Epstein SE, Johnston GS. Sensitivity, specificity and predictive accuracy of radionuclide cineangiography during exercise in patients with coronary artery disease. Comparison with exercise electrocardiography. Circulation. 1979 Sep;60(3):572-80. doi: 10.1161/01.cir.60.3.572. No abstract available. PMID 455620